CLINICAL TRIAL: NCT00843349
Title: Fibroblast Growth Factor-23 Reduction in Predialysis Chronic Kidney Disease
Brief Title: Fibroblast Growth Factor-23 (FGF23) Reduction in Predialysis Chronic Kidney Disease (CKD)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Myles Wolf (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor-Investigator, Myles Wolf, Associate Professor of Medicine, Chief of Division of Nephrology and Hypertension, University of Miami
Organization: University of Miami (Other)
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Prevention
Other Study IDs: 20080536; R01DK076116 (NIH)
Record Dates: First submitted 2009-02-12; First posted 2009-02-13 (Estimated); Results first posted 2013-06-07 (Estimated); Last update posted 2013-06-07 (Estimated); Status verified 2013-05

CONDITIONS: Kidney Disease
Keywords: Phosphorus; Fibroblast Growth Factor-23; Kidney Disease
MeSH Terms: conditions — Kidney Diseases | interventions — lanthanum carbonate

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- 900 mg Phosphate Diet-LC (Active Comparator): dietary phosphorus restriction (900 mg/day of phosphorus) + phosphorus binder (Lanthanum Carbonate)
  Interventions: Drug: Lanthanum Carbonate; Other: 900 mg Phosphate Diet
- Ad Libitum Diet-LC (Active Comparator): no dietary intervention + phosphorus binder (Lanthanum Carbonate)
  Interventions: Drug: Lanthanum Carbonate; Other: Ad Libitum Diet
- 900 mg Phosphate Diet-LC Placebo (Active Comparator): dietary phosphorus restriction (900 mg/day of phosphorus) + placebo
  Interventions: Other: 900 mg Phosphate Diet; Drug: LC Placebo
- Ad Libitum Diet-LC Placebo (Placebo Comparator): no dietary intervention + placebo
  Interventions: Drug: LC Placebo; Other: Ad Libitum Diet

INTERVENTIONS:
Drug: Lanthanum Carbonate — Phosphorus binder
  Other Names: Fosrenol
  Arms: 900 mg Phosphate Diet-LC; Ad Libitum Diet-LC
Other: 900 mg Phosphate Diet — Amount of phosphorus consumption in a day kept below 900 mg.
  Arms: 900 mg Phosphate Diet-LC; 900 mg Phosphate Diet-LC Placebo
Drug: LC Placebo — Placebo for Lanthanum Carbonate
  Other Names: Placebo
  Arms: 900 mg Phosphate Diet-LC Placebo; Ad Libitum Diet-LC Placebo
Other: Ad Libitum Diet — Patients continued to eat their usual diet.
  Arms: Ad Libitum Diet-LC; Ad Libitum Diet-LC Placebo

SUMMARY:
The investigators would like to study the role of phosphorus metabolism in the development of certain hormonal problems in people with chronic kidney disease (CKD). More specifically, the goals of the research are (1) to understand the cause of hyperparathyroidism - a hormone problem that often develops in patients who have kidney disease and (2) to test whether decreasing phosphorus intake could help improve or prevent hyperparathyroidism.

DETAILED DESCRIPTION:
The purposes of this proposal are to (1) develop pilot data of a treatment strategy that manipulates phosphate loading in an effort to ameliorate the development of secondary hyperparathyroidism by increasing endogenous calcitriol levels, which itself, along with decreased phosphate levels, may be potential survival factors; (2) examine the effect of phosphorus restriction/fibroblast growth factor-23 (FGF-23)reduction strategies on insulin resistance and cardiac structure and function in individuals with renal dysfunction. If this proof-of-concept study validates our approach, we will embark on larger trials with extended follow up that would aim to show that the treatment window of phosphate reduction strategies should be expanded to the millions of normophosphatemic patients with early-stage CKD with the ultimate goal being improved survival.

We hypothesize will test the following hypotheses:

1. Decreased dietary phosphorus loading in chronic kidney disease (CKD) patients with normal serum phosphate levels, through dietary restriction, treatment with dietary phosphate binders or a combination of both, will lead to decreased FGF-23 levels, increased calcitriol levels and decreased parathyroid hormone (PTH) levels. In an effort to understand the magnitude and effectiveness of our interventions according to CKD stage, we will test the hypothesis in an equal number of stage 3a (estimated Glomerular Filtration Rate or eGFR 45 - 60 ml/min), stage 3b (eGFR 30 - 45 ml/min) and stage 4 (eGFR 15 - 30 ml/min) CKD patients. This will allow us to define the optimal timing along the spectrum of CKD when our interventions will be most effective which will be critical for planning future longer term outcome studies.
2. Subjects who receive phosphorus reduction strategies will display increased calcitriol levels and decreased insulin resistance from baseline to post-intervention compared to subjects who are randomized to the control arm. The degree of improvement will be modulated such that those who receive both dietary phosphorus restriction and phosphorus binders will display the greatest change.
3. Decreased levels of FGF-23, resulting from phosphorus restriction interventions, will be associated with improved cardiac function, particularly measures of diastolic function as evaluated by pre- and post-intervention echocardiograms.

Overview of Study Design

* Randomized, double-blinded, placebo controlled, physiological, crossover study with a 2 x 2 factorial design of CKD patients
* Written, informed consent will be obtained from all potential subjects at an initial screening visit at the General Clinical Research Center (GCRC), after which they will undergo a brief history and physical, and baseline blood measurements to determine eligibility.
* A certified nutritionist will evaluate subjects' baseline dietary intake during the two week run-in period.
* Eligible subjects will provide two 24-hour urine collections on separate days prior to initiating the protocol to calculate their creatinine clearance and estimate their mean urinary Pi and calcium excretion while eating their usual diets.
* This run-in period will be followed by randomization to binders (Lanthanum Carbonate) vs. placebo and to a phosphorus restricted vs. unrestricted diet
* 25% of subjects will receive binders + restricted diet; 25% binders + unrestricted diet; 25% placebo + restricted diet; and 25% placebo + unrestricted diet (the control group)
* Block randomization will ensure that the 4 intervention groups will include 10 subjects each from CKD stages 3a, 3b and 4 (120 total)
* The nutrition interventions will be managed by a certified nutritionist
* Subjects who are randomized to the unrestricted phosphorus diet arms will be encouraged to maintain their normal eating habits and will not receive any specific dietary counseling from the nutritionist.
* Subjects who are randomized to the phosphorus restriction arms will receive dietary counseling to reduce their phosphorus intake to a target of 900mg/day. If their intake is already estimated to be below that level, they will be encouraged to maintain their current intake. Subjects with lower phosphorus intake at baseline (<900 mg/d) who are randomized to the unrestricted phosphorus diet will not be encouraged to increase their intake.
* All subjects will take a pill, either the phosphorus binder lanthanum carbonate or a placebo, to ensure subject blinding.
* The nutritionist will meet with all subjects regardless of whether they are consuming a reduced phosphate diet or their normal diet. Since it is difficult to reduce phosphorus intake, subjects who are randomized to phosphorus restriction arms will be aware of their intervention. However, subjects who are randomized to the unrestricted phosphorus diet will not be told of their randomization. The nutritionist will counsel them on healthy eating habits as a form of "placebo".
* Three months of follow up post randomization, during which:

  * Fasting blood and urine measures will be repeated every two weeks after randomization throughout the three month intervention. Data for the study endpoints as well as safety data (see below) will be collected at these time points.
  * A certified nutritionist will counsel subjects randomized to the phosphorus restricted diet on how to substitute foods in their diet that are high in phosphorus with foods of equivalent nutritional value that are lower in phosphorus using counseling techniques employed in routine clinical practice. The nutritionist will not advise subjects that are randomized to an unrestricted phosphorus diet to change their eating habits in any way.
  * The nutritionist will use 3-day food records to evaluate the intake of all study subjects over the 3 month intervention. Subjects will receive their first 3-day food record form at the screening visit (visit 1) and return it on visit 2 to be examined by the study nutritionist in preparation for counseling. After the initial counseling session, subjects will bring their completed 3-day food records to the GCRC at visits 4, 7 and 9.
* All subjects will undergo a limited echocardiogram to measure physiological changes in diastolic function pre- and post-intervention.

ELIGIBILITY:
Inclusion Criteria:

* We will include stage 3a, 3b and 4 CKD patients, aged 18 years or over with normal serum phosphate levels (≤ 4.6 mg/dl)

Exclusion Criteria:

* Patients with rapidly advancing renal failure who thus might develop hyperphosphatemia or end stage renal disease requiring initiation of dialysis during the study period
* Patients expected to require dialysis initiation within the follow up period
* Patients with hyperphosphatemia > 4.6 mg/dl
* Patients with any previous or current treatment with phosphate binders or active vitamin D (doxercalciferol or calcitriol)
* Malnutrition, defined as a serum albumin < 3.0 mg/dl
* Patients with liver disease (ALT or AST > 100 U/L) or cholestasis (direct bilirubin > 1.0 mg/dl) because this can limit their ability to absorb fat soluble vitamins such as vitamin D
* Anemia, defined as a hematocrit < 27% at the screening visit
* Medical conditions impacting Pi metabolism-primary hyper- or hypoparathyroidism; Patients with previous subtotal parathyroidectomy; gastrointestinal malabsorption disorders such as Crohn's Disease, ulcerative colitis, celiac disease, or severe liver dysfunction;
* Patients with outpatient counseling by a renal nutritionist within the previous 6 months
* Hospitalization within the previous 4 weeks
* Pregnancy or breastfeeding mothers
* Patients unable to independently provide written informed consent - prisoners, mentally incompetent, minors

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2009-07; Primary Completion 2012-02 (Actual); Study Completion 2012-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Myles Wolf, MD, MMSc, Principal Investigator — University of Miami
Locations (1):
- University of Miami Hospital, Miami, Florida, United States

REFERENCES:
- [Derived] Natale P, Green SC, Ruospo M, Craig JC, Vecchio M, Elder GJ, Strippoli GF. Phosphate binders for preventing and treating chronic kidney disease-mineral and bone disorder (CKD-MBD). Cochrane Database Syst Rev. 2025 Jun 27;6(6):CD006023. doi: 10.1002/14651858.CD006023.pub4. PMID 40576086
- [Derived] Isakova T, Barchi-Chung A, Enfield G, Smith K, Vargas G, Houston J, Xie H, Wahl P, Schiavenato E, Dosch A, Gutierrez OM, Diego J, Lenz O, Contreras G, Mendez A, Weiner RB, Wolf M. Effects of dietary phosphate restriction and phosphate binders on FGF23 levels in CKD. Clin J Am Soc Nephrol. 2013 Jun;8(6):1009-18. doi: 10.2215/CJN.09250912. Epub 2013 Mar 7. PMID 23471131

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants in the study were enrolled between July 2009 and November 2011. Study team members identified potential participants from outpatient clinics at the University of Miami Nephrology Clinics and Jackson Health System Nephrology Clinics.
Pre-assignment Details: After screening, the patients underwent a two-week run-in period encompassing three separate visits during which baseline blood and urine were collected, as well as baseline nutrition information.
Groups:
- 900 mg Phosphate Diet-Lanthanum Carbonate (LC): dietary phosphorus restriction (900 mg/day of phosphorus) + phosphorus binder (Lanthanum Carbonate)
- Ad Libitum Diet-Lanthanum Carbonate: no dietary intervention + phosphorus binder (Lanthanum Carbonate)
- 900 mg Phosphate Diet-Lanthanum Carbonate Placebo: dietary phosphorus restriction (900 mg/day of phosphorus) + Lanthanum Carbonate placebo
- Ad Libitum Diet-Lanthanum Carbonate Placebo: no dietary intervention + Lanthanum Carbonate placebo
Period: Overall Study
Arm/Group | 900 mg Phosphate Diet-Lanthanum Carbonate (LC) | Ad Libitum Diet-Lanthanum Carbonate | 900 mg Phosphate Diet-Lanthanum Carbonate Placebo | Ad Libitum Diet-Lanthanum Carbonate Placebo
Started | 11 | 11 | 10 | 11
Completed | 8 | 11 | 10 | 10
Not Completed | 3 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 900 mg Phosphate Diet-LC | Ad Libitum Diet-LC | 900 mg Phosphate Diet-LC Placebo | Ad Libitum Diet-LC Placebo | Total
Number analyzed (Participants) | 11 | 11 | 10 | 11 | 43
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 10 | 9 | 8 | 9 | 36
  >=65 years | 1 | 2 | 2 | 2 | 7
Age Continuous [Mean (Standard Deviation); unit: years] | 56.1 (10.0) | 55.1 (12.6) | 56.2 (10.1) | 55.1 (12.6) | 55.4 (10.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 3 | 3 | 5 | 14
  Male | 8 | 8 | 7 | 6 | 29
Region of Enrollment [Number; unit: participants]
  United States | 11 | 11 | 10 | 11 | 43

OUTCOME MEASURES:

1. Primary Outcome: Percentage Changes in Fibroblast Growth Factor-23 (FGF-23) Levels
Description: Nonfasting blood was assessed over a period of 12 weeks. The primary endpoint was percentage change in FGF-23 levels from baseline.
Time Frame: Week 0 - 12
Population: All participants that completed their respective intervention periods were selected for analysis.
Measure: Mean (Standard Deviation); unit: percentage of change from baseline
Arm/Group | 900 mg Phosphate Diet-LC | Ad Libitum Diet-LC | 900 mg Phosphate Diet-LC Placebo | Ad Libitum Diet-LC Placebo
Number analyzed (Participants) | 8 | 11 | 10 | 10
percentage of change from baseline | -0.35 (0.32) | 0.25 (0.53) | 0.00 (0.24) | -0.02 (0.29)

2. Primary Outcome: Percentage Changes in Parathyroid Hormone (PTH) Levels
Description: Nonfasting blood was assessed over a period of 12 weeks. Endpoint was percentage changes in PTH levels from baseline.
Time Frame: Week 0 - 12
Population: All participants that completed their respective intervention periods were selected for analysis.
Measure: Mean (Standard Deviation); unit: percentage of change from baseline
Arm/Group | 900 mg Phosphate Diet-LC | Ad Libitum Diet-LC | 900 mg Phosphate Diet-LC Placebo | Ad Libitum Diet-LC Placebo
Number analyzed (Participants) | 8 | 11 | 10 | 10
percentage of change from baseline | 0.04 (0.45) | 0.24 (0.42) | 0.06 (0.22) | 0.17 (0.62)

ADVERSE EVENTS:
Time Frame: Adverse event data was collected all throughout the study, from July 2009 to March 2012.
Arm/Group | 900 mg Phosphate Diet-LC | Ad Libitum Diet-LC | 900 mg Phosphate Diet-LC Placebo | Ad Libitum Diet-LC Placebo
Serious Adverse Events (participants affected / at risk) | 0/11 | 0/11 | 0/10 | 0/11
Other Adverse Events (participants affected / at risk) | 4/11 | 1/11 | 0/10 | 3/11
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 900 mg Phosphate Diet-LC (N=11) | Ad Libitum Diet-LC (N=11) | 900 mg Phosphate Diet-LC Placebo (N=10) | Ad Libitum Diet-LC Placebo (N=11)
Nausea and vomiting (Gastrointestinal disorders) | 3 (3) | 0 (0) | 0 (0) | 2 (2) — Moderate to severe nausea and vomiting
Hypophosphatemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1) — Low serum phosphate levels.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No